CLINICAL TRIAL: NCT01819428
Title: A Prospective, Open-label, Single Arm, Multi-center, Phase II Exploratory Trial to Evaluate the Efficacy and Safety of NOV120101 (Poziotinib) as the First-line Treatment Medication in Patients With Harboring EGFR Mutations
Brief Title: NOV120101 (Poziotinib) for 1st Line Monotherapy in Patients With Lung Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: National OncoVenture (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV120101-201
Record Dates: First submitted 2013-03-14; First posted 2013-03-27 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Adenocarcinoma of Lung Stage IIIB; Adenocarcinoma of Lung Stage IV
Keywords: EGFR mutation; Lung Adenocarcinoma; Firstline therapy; Second generation of tyrosine kinase
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOV120101 (Poziotinib) (Experimental): Single arm study with NOV120101(poziotinib)12mg PO daily administration
  Interventions: Drug: NOV120101 (Poziotinib)

INTERVENTIONS:
Drug: NOV120101 (Poziotinib) — NOV120101 (Poziotinib)12 mg PO once daily until disease progression or unacceptable toxicity development
  Other Names: HM781-36B; Poziotinib

SUMMARY:
The purpose of this open-label, single-arm, multi-center phase II trial is to evaluate the efficacy and safety of novel pan-HER inhibitor, NOV120101 (Poziotinib), as a first-line monotherapeutic agent in patients with lung adenocarcinoma harboring EGFR mutation.

DETAILED DESCRIPTION:
EGFR TKIs are known as more effective and less toxic medications against EGFR mutated tumors. However, newly acquired resistance to these inhibitors is the inevitable obstacle in continuous treatment with them. To overcome this problem, many new class of TKIs including NOV120101 (Poziotinib) are developing these days. To evaluate the efficacy of NOV120101 (Poziotinib) as a first-line monotherapeutic medication, chemotherapy-naïve patients will participate in this study. Subjects will receive NOV120101 (Poziotinib) 12 mg PO once daily until disease progression or unacceptable toxicity development. Objective response rate (ORR) will be analyzed as the primary endpoint in this trial. Secondary endpoints including PFS rate at 12 months, DCR, PFS, and OS will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 20 years or older
2. Pathologically confirmed stage IIIB (unresectable) or IV lung adenocarcinoma
3. Documented EGFR mutation (e.g., exon 19 deletion, exon 21 L858R, etc.) with tumor tissue
4. Patients who have 1 or more measurable lesions according to RECIST version 1.1
5. ECOG performance status 2 or less
6. Life expectancy of 12 weeks or more
7. Patients who have adequate hematological, hepatic and renal functions; WBC 4,000 or more per mm3, platelet 100,000 or more per mm3, serum creatinine 1.5 times or less upper limit of normal, AST and ALT 2.5 times or less upper limit of normal, total bilirubin 1.5 times or less upper limit of normal
8. Patients who give written informed consent voluntarily

Exclusion Criteria:

1. Prior systemic chemotherapy, immunotherapy or biological therapy for stage IIIB or IV adenocarcinoma (However, neo or adjuvant chemo, chemoradio or radiotherapy is permitted if at least 6 months has elapsed prior to disease progression)
2. Prior treatment with small molecules or antibodies targeting EGFR
3. Patients who received major surgery within 4 weeks before study drug administration
4. Symptomatic CNS metastases (patients with radiologically and neurologically stable metastases and being off corticosteroids for at least 2 weeks are able to participate in this trial.)
5. History of other malignancies except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for 3 years or more and considered to be cured by investigator's judgment
6. Known preexisting interstitial lung disease (ILD)
7. NYHA class III or IV heart failure, uncontrolled hypertension, unstable angina or myocardial infarction within 6 months, poorly controlled arrhythmia or other clinically significant cardiovascular abnormalities at investigator's discretion
8. Patients whose left ventricle ejection fraction (LVEF) is below the institutional lower limit of normal (if no lower limit of normal is defined in the site, the lower limit is 50 percent)
9. Patients with known active hepatitis B, HIV infection, or other uncontrolled infectious disease
10. Clinically significant or recent acute gastrointestinal disorders with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption disorders, CTCAE grade 2 diarrhea or more due to any etiology)
11. Patients who cannot receive IP by mouth and be diagnosed with clinically significant gastrointestinal disorders which can prevent administration, transit or absorption of the study drug
12. Pregnancy or breast feeding
13. Women of childbearing potential (WOCBP) or men who are unwilling to use adequate contraception or be abstinent during the trial and for at least 2 months after the end of treatment
14. Patients who received other investigational products except gefitinib and erlotinib within 4 weeks before participation
15. Patients who cannot participate in this trial by investigator's judgment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | about 3 years
  the proportion of patients with complete response (CR) and/or partial response (PR)

SECONDARY OUTCOMES:
Progression free survival (PFS) rate at 12 months | 12 months after enrollment of the last subject
  the proportion of patients with complete response (CR) and/or partial response (PR) at 12 months following start of study drug administration.
Disease control rate (DCR) | 3 years
  the proportion of patients with CR, PR and/or stable disease (SD)
Progression free survival (PFS) | 3 years
  The length of time during and after medication or treatment during which the disease being treated (usually cnacer) does not get worse.
Overall survival (OS) | 3 years
  the time from study drug administration until death from any cause
Change of quality of life (QoL) measured by EQ-5D questionnaire | 3 years
  Change means the end of treatment minus baseline in each patient

OTHER OUTCOMES:
Population pharmacokinetics (PK) of NOV120101 (Poziotinib) | 3 months after enrollment of the last subject
  to observe pharmacokinetic parameter, inter-individual variability and intra-individual variability considering covariates, demographic factors, influencing PK profile.
Subgroup analyses according to the genetic information | 3 years
  to observe HGF expression status in plasma and T790M mutation induction status from plasma DNA

CONTACTS AND LOCATIONS:
Overall Officials: Jungyong Kim, MD, Study Director — National OncoVenture
Locations (6):
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Gachon University Gil Hospital, Namdong-Gu, Incheon
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul
  - Ulsan University Hospital, Dong-gu, Ulsan